CLINICAL TRIAL: NCT00004979
Title: Phase I/II Study of Oral Topotecan and Intravenous Paclitaxel in Patients With Advanced Non-Small Cell Lung Cancer (Phases I and II) and Other Advanced Solid Tumors (Phase I Only)
Brief Title: Topotecan and Paclitaxel in Treating Patients With Advanced Non-small Cell Lung Cancer or Other Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067543; UCLA-9904034; SB-104864/250; NCI-G00-1676
Record Dates: First submitted 2000-03-07; First posted 2004-06-04 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2001-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Paclitaxel; Topotecan

INTERVENTIONS:
Drug: paclitaxel
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining topotecan and paclitaxel in treating patients who have advanced non-small cell lung cancer or other advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: Phase I: I. Determine the maximum tolerated dose (MTD) of oral topotecan combined with a fixed dose of paclitaxel in patients with advanced non-small lung cancer (NSCLC) and other advanced solid tumors. II. Determine the response rate of NSCLC patients treated at the MTD of oral topotecan combined with intravenous paclitaxel. III. Determine the dose limiting toxicities of this drug combination in this patient population. Phase II: IV. Determine the toxicities of this regimen at its MTD in patients with NSCLC. V. Determine time to response, response duration, survival, time to progression, and rate of stable disease of patients with NSCLC treated with this regimen at the MTD. VI. Assess changes in well-being of patients with NSCLC treated with this regimen at the MTD.

OUTLINE: This is a dose escalation study of topotecan. Patients receive oral topotecan on days 1-5 and paclitaxel IV over 3 hours on day 1. Treatment continues every 21 days in the absence of unacceptable toxicity or disease progression. Cohorts of 3-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicities. Once the MTD is determined, additional patients with non-small cell lung cancer are accrued to receive treatment with topotecan and paclitaxel at the recommended phase II dose. Quality of life is assessed in the phase II portion of the study at baseline, before each treatment course, and at the end of the study. Patients are followed at 3 weeks.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for the phase I dose escalation portion of this study. A total of 14-40 additional non-small cell lung cancer patients will be accrued to the phase II portion of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Phase I: Advanced solid tumors, including non-small cell lung cancer (NSCLC), that have failed conventional therapy or for which no standard effective therapy exists May have failed conventional chemotherapy for tumor type Chemotherapy naive NSCLC allowed Measurable or evaluable disease Phase II: Stage IIIB or IV NSCLC not amenable to surgery or radiotherapy with curative intent No prior chemotherapy allowed At least 1 bidimensionally measurable non-CNS indicator lesion defined by diagnostic studies Measurable disease on CT or MRI scan must have one diameter at least 1 cm and one diameter at least 2 cm Measurable disease on chest x-ray must have both diameters at least 2 cm Palpable tumor masses that cannot be evaluated radiologically must have two diameters at least 2 cm Measurable skin lesion must have at least one diameter at least 1 cm and its presence must be evaluated by a photograph At least 6 weeks since prior radiotherapy to measurable, progressive disease No brain and/or leptomeningeal metastases by CT or MRI brain scan unless asymptomatic on neurologic exam and not receiving corticosteroid therapy to control symptoms

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 Life expectancy: At least 12 weeks Hematopoietic: WBC at least 3,000/mm3 Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal SGOT/SGPT no greater than 1.5 times upper limit of normal (ULN) (5 times ULN if liver metastases present) Alkaline phosphatase no greater than 1.5 times ULN (5 times ULN if liver metastases present) Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception for 3 months prior to and during study Able to take oral medication No active infection No other prior or concurrent malignancies except basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix No other severe medical problem unrelated to malignancy that would preclude study compliance or expose patient to extreme risk No condition of the gastrointestinal (GI) tract or otherwise that would affect GI absorption and motility No history of hypersensitivity reactions to paclitaxel or other drugs formulated in polyoxyethylated castor oil

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: See Disease Characteristics No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics Radiotherapy: See Disease Characteristics At least 4 weeks since palliative radiotherapy and recovered No prior radiotherapy to greater than 30% of bone marrow reserve No concurrent radiotherapy Surgery: See Disease Characteristics At least 4 weeks since prior surgery (lesser period acceptable if deemed in best interest of patient) Other: No concurrent metoclopramide or cisapride to maintain motility or gastric emptying At least 30 days or 5 half-lives since other prior investigational drugs for treatment of cancer No other concurrent investigational medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2000-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Figlin, MD, FACP, Study Chair — Jonsson Comprehensive Cancer Center